CLINICAL TRIAL: NCT00758017
Title: Efficacy of Different Acupuncture Methods for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Claudia M. Witt, MD, Institute for Social Medicine, Epidemiology, and Health Economics, Charité
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aku-08
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; acupuncture
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture 1 (Experimental)
  Interventions: Other: Acupuncture 1
- Acupuncture 2 (Active Comparator)
  Interventions: Other: Acupuncture 2

INTERVENTIONS:
Other: Acupuncture 1 — Application of individualised acupuncture
  Arms: Acupuncture 1
Other: Acupuncture 2 — Application of standardised acupuncture
  Arms: Acupuncture 2

SUMMARY:
The aim of the study is to evaluate pain intensity over 8 weeks in acupuncture patients with chronic low back pain and to compare 2 different groups of patients which differ in the acupuncture method used to treat the pain.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic low back pain (for at least 3 months) confirmed by a consultant
* indication for treatment of low back pain with acupuncture confirmed by a consultant
* at least 40 mm on a VAS pain scale

Exclusion Criteria:

* acupuncture during the last 6 months
* start of a new therapy for low back pain within the last 4 weeks
* pregnancy
* substance or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-01; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Pain intensity over 8 weeks (area under the curve) | 8 weeks

SECONDARY OUTCOMES:
Intensity of back pain at week 8 and week 26 | baseline, week 8, week 26
Back function (FFbH-R) | baseline, week 8, week 26
QoL | baseline, week 8, week 26
Days with medication intake | baseline to end of week 8
Days with physical therapy because of back pain | baseline to end of week 8
Sick leave days | baseline, at week 8, at week 26
Number of therapy sessions | baseline to expected time frame 3 months
Duration of therapy | baseline to expected time frame 3 months
Adverse effects and severe adverse effects | baseline to expected time frame 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M. Witt, MD, Principal Investigator — Institute for Social Medicine, Epidemiology, and Health Economics, Charité University Medical Center, Berlin, Germany
Locations (1):
- ambulatory practice Yang-Strobel, Berlin, Germany

REFERENCES:
- [Derived] Pach D, Yang-Strobel X, Ludtke R, Roll S, Icke K, Brinkhaus B, Witt CM. Standardized versus Individualized Acupuncture for Chronic Low Back Pain: A Randomized Controlled Trial. Evid Based Complement Alternat Med. 2013;2013:125937. doi: 10.1155/2013/125937. Epub 2013 Oct 28. PMID 24288556